CLINICAL TRIAL: NCT00003199
Title: A Phase II Trial for Patients With Inflammatory (Stage IIIB) and Responsive Metastatic Stage IV Breast Cancer Using Busulfan, Melphalan and Thiotepa Followed by Autologous or Syngeneic PBSC Rescue and 12 Weeks of Post-Engraftment Immunotherapy With Low-Dose IL-2 and GM-CSF
Brief Title: Combination Chemotherapy and Peripheral Blood Stem Cell Transplant Followed By Aldesleukin and Sargramostim in Treating Patients With Inflammatory Stage IIIB or Metastatic Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 1605; NCI-2010-00728 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Estrogen Receptor-positive Breast Cancer; Inflammatory Breast Cancer; Male Breast Cancer; Progesterone Receptor-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage IIIB Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Breast Neoplasms | interventions — Tamoxifen; Busulfan; Thiotepa; Melphalan; aldesleukin; Interleukin-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Peripheral Blood Stem Cell Transplantation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): See Detailed Description.
  Interventions: Drug: tamoxifen citrate; Drug: busulfan; Drug: thiotepa; Drug: melphalan; Biological: aldesleukin; Biological: sargramostim; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: tamoxifen citrate — Given orally
  Other Names: Nolvadex; TAM; tamoxifen; TMX
Drug: busulfan — Given orally
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: thiotepa — Given IV
  Other Names: Oncotiotepa; STEPA; TESPA; Tespamin; TSPA
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Procedure: peripheral blood stem cell transplantation — Undergo autologous peripheral blood stem cell infusion
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Radiation: radiation therapy — May undergo radiotherapy after completion of IL-2/GM-CSF
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase II trial studies how well giving combination chemotherapy and peripheral blood stem cell transplant followed by aldesleukin and sargramostim works in treating patients with inflammatory stage IIIB or metastatic stage IV breast cancer. Drugs used in chemotherapy, such as busulfan, melphalan, and thiotepa, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. This may allow more chemotherapy to be given so that more tumor cells are killed. Aldesleukin may stimulate the white blood cells to kill breast cancer cells. Giving aldesleukin together with sargramostim may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the event-free survival and survival of patients treated for inflammatory (Stage IIIb) and responsive stage IV breast cancer with BUMELTT and PBSC support and low dose immunotherapy with IL2 and GM-CSF.

SECONDARY OBJECTIVES:

II. To determine the toxicity of a combination of low-dose IL-2 and GM-CSF in patients following HDC with BUMELTT and PBSC support.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive busulfan orally (PO) once every 6 hours on days -8, -7, and -6; melphalan IV over 30 minutes on days -5 and -4; and thiotepa IV over 2 hours on days -3 and -2.

TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell infusion on day 0.

POST-TRANSPLANT THERAPY: All patients receive tamoxifen citrate* PO once daily beginning prior to aldesleukin (IL-2) and sargramostim (GM-CSF) therapy and continuing for 5 years or until relapse (estrogen receptor [ER]- or progesterone receptor [PR]-positive patients) OR until completion of IL-2/GM-CSF therapy (ER-negative or PR-negative patients). Eligible patients receive IL-2 subcutaneously (SC) daily and GM-CSF SC 3 times weekly for 12 weeks beginning 30-100 days after transplantation. Patients may receive radiotherapy after completion of IL-2/GM-CSF treatment if no prior radiotherapy was given before transplantation.

*Stage IV patients not receiving IL-2/GM-CSF therapy who received tamoxifen citrate as part of adjuvant therapy and subsequently failed, receive oral anastrozole once daily for 5 years or until progression instead of tamoxifen.

[*For postmenopausal patients, the choice and duration of hormonal therapy given in addition to or an alternative to tamoxifen therapy will be at the physician's discretion]

Patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory (stage IIIb) or responsive stage IV breast cancer with metastasis to soft tissue and/or bone; responsive stage IV disease is defined as patients who achieve a PR (>= 50% reduction in measurable tumor burden) or CR following initial chemotherapy for metastatic disease or patients with locally recurrent disease (chest wall/axillary nodes) who are rendered disease-free following surgery or radiation therapy without receiving chemotherapy; bone disease is categorized as responsive if there is demonstrated sclerosis of prior lesions with no new lesions
* Patients should have received 4-7 cycles of an Adriamycin and/or taxane-based regimen for stage IIIb or stage IV disease; locally recurrent (chest wall/axillary nodes) patients rendered NED by RT or surgery do not need to receive chemotherapy for stage IV disease prior to Cytoxan/Taxol
* Patient has received Cytoxan 4 gm/m^2 x 1 and Taxol 250 mg/m^2 x 1 per FHCRC protocol 506.03; Cytoxan/Taxol must be given after all other chemotherapy is completed and before transplant
* Stem cells were collected after mobilization with Cytoxan/Taxol or after mobilization from an FHCRC approved cytokine protocol; if syngeneic collection, PBSC's were collected by using G-CSF according to FHCRC protocol 753; patient has an adequate number of peripheral blood stem cells stored (>= 2.5 x 10^6 CD34+ cells/kg)
* The patient must have the capacity to give informed consent; the patient must have signed an approved consent form conforming with federal and institutional guidelines
* Hepatic function: Bilirubin =< 2 mg%; SGOT or SGPT =< 2.5 x institutional normal
* Renal function: Creatinine =< 2.0 mg/dl or a creatinine clearance >= 50 mg/min
* Pre-Study tests have been performed as outlined in the Study Calendar
* Patients will begin IL-2/GM-CSF therapy if they meet the following criteria post-transplant:
* Can start therapy 30 to 100 days after transplant
* Karnofsky performance status > 60
* ANC > 1,000 cells/mm^3 and platelets > 30,000/cells/mm^3 (transfusion independent) for at least 5 days before starting therapy
* Total bilirubin =< 2.5 x upper limit of normal
* SGOT =< 2.5 x upper limit of normal
* Creatinine =< 2.0 mg/dl

Exclusion Criteria:

* Patients with a Karnofsky Performance Score less than 70
* Patients with a left ventricular ejection fraction less than 50 % (LVEF must be performed in patients with symptoms of CHF, abnormal cardiac exam or history of Adriamycin therapy total dose > 400 mg/m^2)
* Patient is pregnant
* Patient is seropositive for the human immunodeficiency virus
* Patients with a history of seizures
* Patients with hypersensitivity to E.coli preparations
* Patients with active auto-immune disease
* Patients with clinically significant pulmonary disease, i.e., diffusion capacity corrected < 60% of predicted; patients with pulmonary problems should be evaluated with appropriate pulmonary studies and/or consult
* Patients with a history of CNS lesion (brain or carcinoid meningitis)
* Patients with significant active infection precluding transplant
* Patients who have had more than one prior chemotherapy regimen for stage IV disease or a prior transplant for any stage disease
* Patients who have had CD34+ selection of their PBSC products
* Patients will not receive IL-2/GM-CSF therapy if they:
* Are > 100 days from transplant
* Have documented disease progression after transplant
* Have an active infection
* Manifested cardiac complications during the initial transplant period, including arrhythmias (that required therapy), congestive heart failure, angina, myocardial infarct, or decreased LVEF to < 45%
* Currently have pericardial effusions, pleural effusions or ascites
* Manifested pulmonary toxicity during the initial transplant period and have a diffusion capacity corrected =< 60%
* Are on steroids
* Currently have a Grade 3 toxicity from BuMelTT
* If the patient does not wish to receive the therapy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1997-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/Puget Sound Oncology Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer: See Detailed Description.
  tamoxifen citrate: Given orally
  busulfan: Given orally
  thiotepa: Given IV
  melphalan: Given IV
  aldesleukin: Given SC
  sargramostim: Given SC
  peripheral blood stem cell transplantation: Undergo autologous peripheral blood stem cell infusion
  radiation therapy: May undergo radiotherapy after completion of IL-2/GM-CSF
Period: Overall Study
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
Started | 50
Completed | 28
Not Completed | 22
Not completed — Refused Post-Transplant Immunotherapy | 5
Not completed — Lack of insurance clearance | 2
Not completed — Screen fail | 15

BASELINE CHARACTERISTICS:
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival of patients treated for inflammatory (Stage IIIb) and responsive stage IV breast cancer with BUMELTT and PBSC support and low dose immunotherapy with IL2 and GM-CSF.
Time Frame: 11 years
Population: Study-wide, 20 patients out of 50 have event-free survival.
Measure: Count of Participants; unit: Participants
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
Number analyzed (Participants) | 50
Participants
  Stage IIIB Disease: number analyzed (Participants) | 18
  Stage IIIB Disease | 11
  Stage IV Disease: number analyzed (Participants) | 32
  Stage IV Disease | 9

2. Secondary Outcome: Overall Survival
Description: Overall survival of patients treated for inflammatory (Stage IIIb) and responsive stage IV breast cancer with BUMELTT and PBSC support and low dose immunotherapy with IL2 and GM-CSF.
Time Frame: 11 years
Measure: Count of Participants; unit: Participants
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
Number analyzed (Participants) | 50
Participants | 18

3. Secondary Outcome: Number of Participants With Toxicity of a Combination of Low-dose IL-2 and GM-CSF
Description: IL-2/GM-CSF toxicity assessed using the NCI Toxicity Criteria. Toxicity was defined as any grade 2, 3, 4 or 5 CNS (except grade 0-3 malaise and fatigue) toxicity; any grade 3, 4, or 5 non-CNS or non-hematological toxicity (except grade 0-3 bilirubin); or any grade 4 or 5 hematological toxicity.
Time Frame: 16 Weeks
Population: 28 (56%) of 50 patients started IL-2/GM-CSF immunotherapy. Stopping rules were not met for this study.
Measure: Count of Participants; unit: Participants
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
Number analyzed (Participants) | 28
Participants | 6

ADVERSE EVENTS:
Time Frame: BUMELTT toxicity assessed day -8 through day 100 using the Bearman Toxicity Criteria, Grades 3 and 4. IL-2/GM-CSF toxicity over 16 weeks will be assessed using the NCI Toxicity Criteria, Grades 3 and 4.
Arm/Group | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer
All-Cause Mortality (participants affected / at risk) | 32/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer (N=50)
Prolonged hospitalization for post-transplant complications (Infections and infestations) | 1 — Transplant toxicity.
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 1 — IL-2/GM-CSF toxicity.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | TX/Maintenance Therapy for Stage IIIB/IV Breast Cancer (N=50)
Myelosuppression (Blood and lymphatic system disorders) | 50 — Toxicity to transplant therapy. No deaths in 1st 100 days post-transplant.
Infections (Infections and infestations) | 16 — Toxicity to transplant therapy. No deaths in 1st 100 days post-transplant.
Hematologic (Blood and lymphatic system disorders) | 6/28 — Toxicity to IL-2/GM-CSF Therapy. No deaths on therapy.
Infection (Infections and infestations) | 3/28 — Toxicity to IL-2/GM-CSF Therapy. No deaths on therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No